CLINICAL TRIAL: NCT05462756
Title: A Phase 3, Parallel-Design, Open-Label, Randomized Controlled Study to Evaluate the Efficacy and Safety of LY3209590 as a Weekly Basal Insulin Compared to Insulin Glargine in Adults With Type 2 Diabetes on Multiple Daily Injections
Brief Title: A Study of Insulin Efsitora Alfa (LY3209590) as a Weekly Basal Insulin Compared to Insulin Glargine in Adult Participants With Type 2 Diabetes on Multiple Daily Injections
Acronym: QWINT-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18260; I8H-MC-BDCV (Other: Eli Lilly and Company); 2021-005878-25 (EudraCT Number)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes; Type 2 Diabetes Treated With Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 500 U/mL - Insulin Efsitora (Experimental): Participants received 500 units per milliliter (U/mL) Insulin Efsitora Alfa (insulin efsitora) administered subcutaneously (SC) once weekly (QW) along with 100 U/mL insulin lispro given SC with meals as needed.
  Interventions: Drug: Insulin Efsitora Alfa; Drug: Insulin Lispro (U100)
- 100 U/mL - Insulin Glargine (Active Comparator): Participants received 100 U/mL insulin glargine administered SC once daily (QD) along with 100 U/mL insulin lispro given SC with meals as needed.
  Interventions: Drug: Insulin Lispro (U100); Drug: Insulin Glargine (U100)

INTERVENTIONS:
Drug: Insulin Efsitora Alfa — Administered SC
  Other Names: LY3209590 and Basal Insulin-FC
  Arms: 500 U/mL - Insulin Efsitora
Drug: Insulin Lispro (U100) — Administered SC
  Other Names: Humalog
Drug: Insulin Glargine (U100) — Administered SC
  Other Names: Basaglar
  Arms: 100 U/mL - Insulin Glargine

SUMMARY:
The reason for this study is to evaluate if the once-weekly study drug insulin efsitora alfa (LY3209590) is safe and effective compared with daily insulin glargine in participants with Type 2 diabetes (T2D) that have already been treated with basal insulin and at least 2 injections per day of prandial insulin. The study consists of a 3-week screening/lead-in period, a 26-week treatment period and a 5-week safety follow-up period. The study will last up to 34 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of T2D according to the world health organization (WHO) criteria, currently treated with basal insulin and at least 2 injections of prandial insulin per day.
* Are receiving ≥10 units of total basal insulin per day at screening.
* Are receiving ≤2 units/kilogram/day of total daily insulin at screening
* Have an HbA1c value of 7.0% to 10%, inclusive, as determined by the central laboratory at screening
* Have been treated with a stable regimen of one of the following basal insulins used according to local product label with or without noninsulin diabetes therapy for at least 90 days prior to screening

  * once daily U-100 or U-200 insulin degludec
  * once daily U-100 or U-300 insulin glargine
  * once or twice daily U-100 insulin detemir or
  * once or twice daily human insulin Neutral Protamine Hagedorn
* Have been treated with at least twice daily dosing of one of the following insulins used according to local product label for at least 90 days prior to screening. One dose of prandial insulin must occur at the evening meal.

  * Insulin lispro-aabc
  * Insulin lispro (U-100 and U-200)s, IN], U-100 or U200)
  * Insulin aspart (U-100)
  * Insulin glulisine (U-100), or
  * Regular insulin (U-100)
* Acceptable noninsulin diabetes therapies may include 0 to up to 3 of the following with a stable dose for at least 90 days prior to screening

  * dipeptidyl peptidase IV inhibitors
  * sodium-glucose co-transporter-2 inhibitors
  * biguanides (for example, metformin), or
  * glucagon-like peptide-1 receptor agonists Note: All noninsulin diabetes therapies must be used in accordance with the corresponding local product label at the time of screening, and participants should be willing to continue stable dosing throughout the study
  * Have a body mass index ≤45 kilogram/square meter (kg/m²)

Exclusion Criteria:

* Have a diagnosis of type 1 diabetes mellitus or latent autoimmune diabetes, or specific type of diabetes other than T2D (for example, monogenic diabetes, diseases of the exocrine pancreas, drug-induced or chemical-induced diabetes).
* Are currently receiving any of the following insulin therapies anytime in the past 90 days:

  * insulin mixtures
  * insulin human, inhalation powder, or
  * continuous subcutaneous insulin infusion therapy, or
  * regular insulin U-500
* Have a history of greater than 1 episode of ketoacidosis or hyperosmolar state/coma requiring hospitalization in the 6 months prior to screening
* Have had any episodes of severe hypoglycemia, defined as requiring assistance due to neurologically disabling hypoglycemia, within the 6 months prior to screening
* Have hypoglycemia unawareness in the opinion of the investigator
* Anticipate making changes in personal CGM or flash glucose monitoring (FGM) use (for example, initiation, stopping, or changing device) during the study.
* Have had New York Heart Association Class IV heart failure or any of the following cardiovascular conditions in the past 3 months prior to screening: acute myocardial infarction, cerebrovascular accident (stroke), or coronary bypass surgery.
* Have undergone gastric bypass (bariatric) surgery, restrictive bariatric surgery, or sleeve gastrectomy within 1 year prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) Mon- Fri 9 AM -5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (80):
- United States (23):
  - CMR of Greater New Haven, LLC, Hamden, Connecticut
  - Tampa Bay Medical Research, Clearwater, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Encore Medical Research - Weston, Weston, Florida
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Research Foundation of SUNY - University of Buffalo, Buffalo, New York
  - Remington Davis Clinical Research, Columbus, Ohio
  - Aventiv Research, Dublin, Ohio
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Research Institute of Dallas, Plano, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Rainier Clinical Research Center, Renton, Washington
- Argentina (16):
  - CEDIC, CABA, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Mautalen Salud e Investigación, Buenos Aires, Buenos Aires F.D.
  - CIPREC, CABA, Buenos Aires F.D.
  - Consultorio de Investigación Clínica EMO SRL, Ciudad Autonoma de Buenos Aire, Buenos Air
  - Instituto Centenario, CABA, Ciudad Autónoma de Buenos Aire
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Ciudad Autonoma de Buenos Aire, Ciudad Autónoma de Buenos Aire
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
  - Centro de Salud e Investigaciones Médicas, Santa Rosa, La Pampa Province
  - Instituto de Investigaciones Clinicas Rosario-Sanatorio Delta, Rosario, Santa Fe Province
  - Instituto Médico Catamarca IMEC, Rosario, Santa Fe Province
  - Centro de Investigaciones Médicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - CENUDIAB, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro de Investigaciones Clinicas del Litoral, Santa Fe
- Germany (7):
  - ClinPhenomics GmbH & Co KG, Frankfurt am Main, Hesse
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - Schwerpunktpraxis für Diabetes und Ernährungsmedizin Dr. med. Winfried Keuthage, Münster, North Rhine-Westphalia
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Diabetespraxis Mergentheim, Bad Mergentheim
  - Diabeteszentrum Hamburg West, Hamburg
- India (6):
  - Life Care Hospital and Research Centre, Bangalore, Karnataka
  - Topiwala National Medical College & B. Y. L. Nair Charitable Hospital, Mumbai, Maharashtra
  - BSES MG Hospital, Mumbai, Maharashtra
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Osmania General Hospital, Hyderabad, Telangana
  - Post Graduate Institute of Medical Education & Research (PGIMER), Chandigarh
- Italy (8):
  - Osepdale Civile Fr 5, Ceccano, Frosinone
  - "Fatebenefratelli Isola Tiberina - Gemelli Isola", Rome, Lazio
  - Ospedale san Giovanni di Dio-Diabetologia, Olbia, Sardinia
  - INRCA Ancona, Ancona
  - IRCCS - AOU di Bologna, Bologna
  - Azienda Ospedaliera Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - Azienda di Rilievo Nazionale e Alta Specializzazione Civico Di Cristina Benfratelli, Palermo
- Mexico (6):
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara, Jalisco
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Unidad Médica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, S.C., Ciudad Madero, Tamaulipas
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
- Puerto Rico (2):
  - Centro de Endocrinologia Alcantara Gonzalez, Bayamón
  - Manati Center for Clinical Research, Manatí
- Spain (12):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol, A Coruña [La Coruña]
  - Hospital Universitario Virgen de la Victoria, Málaga, Andalusia
  - Hospital Universitari Son Espases, Palma, Balears [Baleares]
  - Hospital Clínico Universitario de Valladolid, Valladolid, Castille and León
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Vithas Hospital Sevilla, Seville, Sevilla
  - Hospital Universitario de La Ribera, Alzira, Valenciana, Comunitat
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario San Cecilio, Granada
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Miller E, Davidson MB, Bajaj HS, Rosenstock J, Philis-Tsimikis A, Bergenstal RM, Case M, Ilag L, Threlkeld R, Levasseur E, Gelsey F. Evaluation of Overall Health State, Treatment Burden, and Satisfaction with Insulin Efsitora Alfa (Efsitora) vs. Daily Comparator in Adults with Type 2 Diabetes in the QWINT Clinical Trial Program. Diabetes Ther. 2026 Jan 27. doi: 10.1007/s13300-025-01833-5. Online ahead of print. PMID 41591636
- [Derived] Blevins T, Dahl D, Perez Manghi FC, Murthy S, Ortiz Carrasquillo R, Li X, Chang AM, Carr MC, Katz M. Once-weekly insulin efsitora alfa versus once-daily insulin glargine U100 in adults with type 2 diabetes treated with basal and prandial insulin (QWINT-4): a phase 3, randomised, non-inferiority trial. Lancet. 2025 Jun 28;405(10497):2290-2301. doi: 10.1016/S0140-6736(25)01069-4. Epub 2025 Jun 22. PMID 40562048
- See also: A Study of LY3209590 as a Weekly Basal Insulin Compared to Insulin Glargine in Adult Participants With Type 2 Diabetes on Multiple Daily Injections (QWINT-4) — https://trials.lilly.com/en-US/trial/350915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants underwent a 26-week treatment period, followed by a 5-week safety follow-up period.
Groups:
- 500 U/mL - Insulin Efsitora: Participants received 500 units per milliliter (U/mL) Insulin Efsitora Alfa (insulin efsitora) administered subcutaneously (SC) once weekly (QW) along with 100 U/mL insulin lispro given SC.
- 100 U/mL - Insulin Glargine: Participants received 100 U/mL insulin glargine administered SC once daily (QD) along with 100 U/mL insulin lispro given SC.
Period: Treatment Period
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Started | 365 | 365
Received At Least 1 Dose of Study Drug | 365 | 365
Completed | 348 | 344
Not Completed | 17 | 21
Not completed — Adverse Event | 3 | 0
Not completed — Assigned Treatment by Mistake | 4 | 3
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Non-Compliance with Study Drug | 1 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 5 | 12
Period: Follow-Up Period
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Started | 357 (Per statistical analysis plan, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.) | 354 (Per statistical analysis plan, participants who completed the study treatment period were required to complete a safety follow-up period and participants who discontinued the study treatment prematurely were encouraged to remain in the study for safety monitoring.)
Completed | 352 | 349
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 0 | 4

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- 500 U/mL - Insulin Efsitora: Participants received 500 U/mL insulin efsitora administered SC QW along with 100 U/mL insulin lispro given SC.
- 100 U/mL - Insulin Glargine: Participants received 100 U/mL insulin glargine administered SC QD along with 100 U/mL insulin lispro given SC.
- Total: Total of all reporting groups
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine | Total
Number analyzed (Participants) | 365 | 365 | 730
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (10.5) | 59.4 (10.5) | 58.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 193 | 176 | 369
  Male | 172 | 189 | 361
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 201 | 203 | 404
  Not Hispanic or Latino | 163 | 161 | 324
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 46 | 45 | 91
  Asian | 54 | 51 | 105
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 11 | 31
  White | 245 | 258 | 503
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 83 | 83 | 166
  Germany | 27 | 24 | 51
  India | 50 | 50 | 100
  Italy | 11 | 15 | 26
  Mexico | 85 | 84 | 169
  Spain | 35 | 35 | 70
  United States | 74 | 74 | 148
HemoglobinA1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Population: All participants who received at least one dose of study drug and had baseline HbA1c value.
  Percentage of HbA1c
    number analyzed (Participants) | 361 | 362 | 723
    (all) | 8.17 (0.83) | 8.18 (0.79) | 8.18 (0.81)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) [Noninferiority]
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time.
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug and had at least one post-baseline HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 361 | 362
Percentage of HbA1c | -1.01 (0.0463) | -1.00 (0.0463)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; Least Squares (LS) Mean was determined using ANCOVA model with Baseline + Country + Personal Use of CGM or FGM at Randomization + Treatment (Type III sum of squares) as variables. Missing data at Week 26 were imputed by return-to-baseline multiple imputations approach. A total of 100 datasets were imputed; Test type: Non-Inferiority — The sample size provided >99% statistical power to show noninferiority assuming a 0.4% noninferiority margin (NIM), in insulin efsitora doses compared to insulin glargine, in a 1:1 randomization, a standard deviation (SD) of 1.1%, and a dropout rate of 15%; LS Mean Difference = -0.012, 95% CI 2-sided [-0.140 to 0.116]

2. Secondary Outcome: Change From Baseline in HbA1c [Superiority]
Description: as for outcome 1
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug and had at least one post-baseline HbA1c data.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 361 | 362
Percentage of HbA1c | -1.01 (0.0463) | -1.00 (0.0463)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.855, ANCOVA; LS Mean Difference = -0.012, 95% CI 2-sided [-0.140 to 0.116]

3. Secondary Outcome: Percentage of Participants Achieving HbA1c <7% Without Nocturnal Hypoglycemia
Description: Percentage of participants achieving HbA1c <7% without nocturnal hypoglycemia [<54 milligram/deciliter (mg/dL) 3.0 millimole/Liter (mmol/L)] or severe during treatment phase up to week 26. Nocturnal hypoglycemia is a hypoglycemia event, including severe hypoglycemia, that occurs at night and presumably during sleep between midnight and 6:00 am.
Time Frame: Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Number; unit: Percentage of participants
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 361 | 362
Percentage of participants | 38.6 | 35.9
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; Test type: Superiority; p = 0.504, Chi-squared; Odds Ratio (OR) = 1.11, 95% CI 2-sided [0.81 to 1.52]

4. Secondary Outcome: Nocturnal Hypoglycemia Event Rate
Description: The event rate of participant-reported clinically significant nocturnal hypoglycemia, (where glucose <54 mg/dL (3.0 mmol/L) or severe and occurs at night and presumably during sleep between midnight and 6:00 AM), measured during treatment phase up to week 26. Group mean is reported here.
Time Frame: Baseline Up To Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 365 | 365
Events per year | 0.67 (0.112) | 1.00 (0.151)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; Group mean is determined by Negative Binomial Model using Number of episodes = Baseline hypoglycemia rate + Hemoglobin A1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as an offset variable; Test type: Superiority; p = 0.058, Negative binomial model; Relative rate = 0.67, 95% CI 2-sided [0.44 to 1.01] — Relative rate is the ratio of the group means (Insulin Efsitora vs Insulin Glargine)

5. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Change from baseline in fasting glucose measured by self-monitoring blood glucose (SMBG).
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 361 | 361
milligrams per deciliter (mg/dL) | -30.87 (1.876) | -26.58 (1.871)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined using ANCOVA model using Baseline + Country + Personal Use of CGM or FGM at Randomization + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at Week 26 were imputed by return-to-baseline multiple imputations approach. A total of 100 datasets were imputed with one for each of the 100 datasets imputed at Baseline; Test type: Superiority; p = 0.104, ANCOVA; LS Mean Difference = -4.29, 95% CI 2-sided [-9.461 to 0.886]

6. Secondary Outcome: Percentage of Time in Glucose Range
Description: Percentage of Time in glucose range between 70 and 180 mg/dL (3.9 and 10.0 mmol/L), inclusive measured during the continuous glucose monitoring (CGM) session.
Time Frame: Week 22 to Week 26
Population: All participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 359 | 360
Percentage of time | 58.39 (0.993) | 57.05 (0.990)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined using ANCOVA model using Baseline + Country + Personal Use of CGM or FGM at Randomization + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at Week 22-Week 26 were imputed by return-to-baseline multiple imputations approach. A total of 100 datasets were imputed with one for each of the 100 datasets imputed at Baseline; Test type: Superiority; p = 0.337, ANCOVA; LS Mean Difference = 1.35, 95% CI 2-sided [-1.404 to 4.101]

7. Secondary Outcome: Percentage of Time in Hypoglycemia Range
Description: Percentage of Time in hypoglycemia range with glucose <54 mg/dL (3.0 mmol/L), measured by CGM.
Time Frame: Week 22 to Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 359 | 360
Percentage of time | 6.84 (0.700) | 5.25 (0.680)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by ANCOVA model using Baseline + Country + Personal Use of CGM or FGM at Randomization + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares) as variables. Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at Week 22-Week 26 were imputed by return-to-baseline multiple imputations approach. A total of 100 datasets were imputed with one for each of the 100 datasets imputed at Baseline; Test type: Superiority; p = 0.104, ANCOVA; LS Mean Difference = 1.59, 95% CI 2-sided [-0.327 to 3.508]

8. Secondary Outcome: Percentage of Time in Hyperglycemia Range
Description: Percentage of Time in hyperglycemia range with glucose >180 mg/dL (10.0 mmol/L), measured by CGM.
Time Frame: Week 22 to Week 26
Population: All participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Percentage of time
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 359 | 360
Percentage of time | 40.10 (1.024) | 41.60 (1.024)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by ANCOVA model using Baseline + Country + Personal Use of CGM or FGM at Randomization + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares). Missing data at Baseline were imputed with multiple imputation with assumption of missing at random. Missing data at Week 22-Week 26 were imputed by return-to-baseline multiple imputations approach. A total of 100 datasets were imputed with one for each of the 100 datasets imputed at Baseline; Test type: Superiority; p = 0.304, ANCOVA; LS Mean Difference = -1.50, 95% CI 2-sided [-4.358 to 1.360]

9. Secondary Outcome: Glucose Variability Between Weeks 22 to 26
Description: Glucose variability measured as coefficient of variation for glucose within day for 24-hour period between Week 22 and 26 was reported.
Time Frame: Week 22 to Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Coefficient of Variation
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 334 | 341
Coefficient of Variation | 28.51 (0.259) | 28.28 (0.254)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by MMRM model with BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Personal Use CGM or FGM at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Unstructured variance-covariance structure was used; Test type: Superiority; p = 0.523, Mixed Models Analysis; LS Mean Difference = 0.23, 95% CI 2-sided [-0.48 to 0.95]

10. Secondary Outcome: Basal Insulin Dose at Week 26
Description: Average weekly basal Insulin Dose at Week 26 was reported.
Time Frame: Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Units per week of basal insulin
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 360 | 362
Units per week of basal insulin | 391.59 (7.482) | 426.62 (7.323)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by Mixed Model Repeated Measures (MMRM) model using BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Personal Use CGM or FGM at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -35.04, 95% CI 2-sided [-55.57 to -14.50]

11. Secondary Outcome: Bolus Insulin Dose at Week 26
Description: Average daily bolus Insulin Dose at Week 26 was reported.
Time Frame: Week 26
Population: All participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Units per day of bolus insulin
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 275 | 285
Units per day of bolus insulin | 27.01 (1.182) | 34.56 (1.156)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by MMRM model using BASELINE + Hemoglobin A1c Stratum at Baseline + Country + Personal Use CGM or FGM at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares) as variables. Variance-covariance structure was set as compound symmetry; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -7.55, 95% CI 2-sided [-10.79 to -4.30]

12. Secondary Outcome: Total Insulin Dose at Week 26
Description: Average total weekly insulin dose at Week 26 was reported.
Time Frame: Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Units per week of insulin
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 274 | 285
Units per week of insulin | 592.92 (12.560) | 666.43 (12.144)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -73.50, 95% CI 2-sided [-107.81 to -39.20]

13. Secondary Outcome: Basal Insulin Dose to Total Insulin Dose Ratio at Week 26
Description: Basal insulin dose to total insulin dose ratio at Week 26 was reported.
Time Frame: Week 26
Population: All participants who received at least one dose of the study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 274 | 285
Ratio | 70.09 (0.749) | 66.55 (0.722)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = 3.53, 95% CI 2-sided [1.49 to 5.58]

14. Secondary Outcome: Hypoglycemia Event Rate
Description: Hypoglycemia event rate was reported. Hypoglycemia with glucose <54 mg/dL (Level 2) or Severe Hypoglycemia (Level 3) was reported. A severe hypoglycemic event is characterized by altered mental or physical status requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions for the treatment of hypoglycemia. Group mean was reported here.
Time Frame: Baseline up to Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Mean (Standard Error); unit: Events per year
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 365 | 365
Events per year | 6.58 (0.709) | 5.94 (0.618)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; Group mean was reported and determined by Negative binomial method using Baseline hypoglycemia rate + Hemoglobin A1c at Baseline (%) + Treatment, with log (exposure in days/365.25) as variables; Test type: Superiority; p = 0.442, Negative binomial model; Mean Difference (Net) = 1.11, 95% CI 2-sided [0.85 to 1.44]

15. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was reported.
Time Frame: Baseline, Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 365 | 363
kilograms (kg) | 2.67 (0.165) | 2.53 (0.165)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by MMRM model using BASELINE + Treatment + Time + Treatment*Time (Type III sum of squares) as variables; Test type: Superiority; p = 0.543, Mixed Models Analysis; LS Mean Difference = 0.14, 95% CI 2-sided [-0.32 to 0.60]

16. Secondary Outcome: Treatment Experience for Diabetes Injection Device at Week 26 - Experience Questionnaire (DID-EQ)
Description: The DID-EQ is a self-administered, 10-item questionnaire designed to assess participants' perceptions of diabetes injection delivery systems for diabetes. The Device Characteristic Subscale is comprised of items 1 to 7 which focus on specific characteristics of injection devices. Each item is rated on a four-point Likert scale. Scores are transformed and range from 0 to 100. Higher scores indicate more positive perceptions of injection device characteristics
Time Frame: Week 26
Population: All participants who received at least one dose of study drug and had evaluable data for this outcome.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
Number analyzed (Participants) | 274 | 286
Score on a scale | 88.1 (0.77) | 86.3 (0.75)
Statistical Analysis 1: Comparison: 500 U/mL - Insulin Efsitora vs 100 U/mL - Insulin Glargine; LS Mean was determined by ANCOVA model using Country + Personal Use CGM or FGM at Randomization + Hemoglobin A1c Stratum at Baseline + Treatment (Type III sum of squares) as variables; Test type: Superiority; p = 0.099, ANCOVA; LS Mean Difference = 1.8, 95% CI 2-sided [-0.3 to 4.0]

ADVERSE EVENTS:
Time Frame: Baseline Through Safety Follow-Up (Up To 31 Weeks)
Description: All participants who received at least one dose of the study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly. Based on the planned safety analysis, adverse event analysis was planned as per the cohorts corresponding to the actual regimen received.
Arm/Group | 500 U/mL - Insulin Efsitora | 100 U/mL - Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 1/365 | 1/365
Serious Adverse Events (participants affected / at risk) | 25/365 | 24/365
Other Adverse Events (participants affected / at risk) | 35/365 | 40/365
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 500 U/mL - Insulin Efsitora (N=365) | 100 U/mL - Insulin Glargine (N=365)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (3) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Spinal instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/193 (1) | 0/176 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Acute psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Postrenal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 U/mL - Insulin Efsitora (N=365) | 100 U/mL - Insulin Glargine (N=365)
Influenza (Infections and infestations) | 14 (17) | 19 (20)
Nasopharyngitis (Infections and infestations) | 23 (25) | 21 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT05462756/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT05462756/SAP_001.pdf